CLINICAL TRIAL: NCT03317314
Title: Cardiopulmonary Interactions in Patients With Heart Failure (Kardio-pulmonale Interaktionen Bei Patienten Mit Linksherzerkrankungen)
Brief Title: Cardiopulmonary Interactions in Patients With Heart Failure
Status: Withdrawn | Type: Observational
Why Stopped: Study was considered not useful and competing with another study in clinical context
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Karen Olsson, PD Dr., PD Dr. med. Karen Olsson, Hannover Medical School
Other Study IDs: Nr. 7155
Record Dates: First submitted 2017-07-05; First posted 2017-10-23 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Heart Failure; Pulmonary Hypertension; Heart Failure With Reduced Ejection Fraction; Heart Failure With Normal Ejection Fraction
MeSH Terms: conditions — Heart Failure; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10 ml samples each for storing plasma and serum samples (biobanking)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Lung Biopsy during LVAD Implantation — Lung Biopsy during LVAD Implantation

SUMMARY:
This study aims to evaluate cardiopulmonary interactions in patients with heat failure

DETAILED DESCRIPTION:
Heart failure is one of the most common diseases, especially in ageing populations, affecting ≥10% of persons 70 years of age or older. There is a growing body of evidence that dyspnea in patients with heart failure is not only related to low cardiac output and pulmonary venous congestion, but also to functional and structural alterations of the lungs.Pulmonary hypertension is a well-known complication of heart failure, but recent evidence suggests that the alveolo-capillary membrane is also affected, at least in subgroups of patients with heart failure.

Damage to the alveolo-capillary membrane is reflected by a low diffusion capacity of the lungs for carbon monoxide (DLCO).

In this study we aim to describe the alteration of lung function and obtain morphometric data of the capillary bed of patients with heart failure.

ELIGIBILITY:
Inclusion criteria

* Written informed consent prior to initiation of any study-mandated procedures
* Male or female ≥40 years at screening
* Confirmed diagnosis of HFpEF (Heart failure with preserved ejection fraction), HFmrEF (heart failure with mid range ejection fraction) or HFrEF (Heart failure with reduced ejection fraction) in New York Heart Association (NYHA) Functional Class II, III or IV

Exclusion criteria

* Significant lung disease according to the judgment of the investigator; as a rule, the total lung capacity (TLC) should be >70% of the predicted value and the forced expiratory volume in 1 second (FEV1) should be >60% of the predicted value
* Significant co-morbidities expected to limit life expectancy to less than 2 years, according to the judgment of the investigator

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients with heart failure ≥40 years at screening.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function in Heart failure | Every Year up tp 36 months
  Pulmonary Function including DLCO (diffusion capacity of the lungs for carbon monoxide)
Relationship DLCO and hemodynamics | Every year up to 36 months, hemodynamics are not mandatory
  To study the relationship between DLCO, KCO (diffusion capacity per unit alveolar volume) and hemodynamics in patients with heart failure
Risk factors for a low DLCO | Baseline, Phone visit every 6 months up to 36 months
  Obtain risk factors for a low DLCO
Impact of LVAD (left ventricular assist device) implantation on lung function | LVAD implantation, 6 months after LVAD implantation, LVAD explantation, 6 months after LVAD explantation, and yearly up to 36 months
  Impact of LVAD implantation on lung function
Predictors of survival and heart-failure related hospitalisations | Baseline, 1 year, Phone visit every 6 months, up to 36 months
  Predictors of survival and heart-failure related hospitalisations

SECONDARY OUTCOMES:
Morphometric data of the pulmonary capillary bed | Biopsies are taken once during LVAD implantation, Heart transplantation or LVAD explantation if performed (variable time points) and compared with the functional assessments, in particular with DLCO and KCO up to 36 months.
  1. To obtain morphometric data on the pulmonary microvasculature in patients with heart failure by taking open lung biopsies from patients with heart failure undergoing heart transplantation or LVAD implantation. The morphometric data will be compared with the functional assessments, in particular with DLCO and KCO.

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Olsson, PD Dr. med., Principal Investigator — Hannover MS
Locations (1):
- Hannover MS, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoeper MM, Meyer K, Rademacher J, Fuge J, Welte T, Olsson KM. Diffusion Capacity and Mortality in Patients With Pulmonary Hypertension Due to Heart Failure With Preserved Ejection Fraction. JACC Heart Fail. 2016 Jun;4(6):441-9. doi: 10.1016/j.jchf.2015.12.016. Epub 2016 Feb 10. PMID 26874383